CLINICAL TRIAL: NCT02211690
Title: The Tolerability of, and Adherence to, Dolutegravir With Co-formulated Tenofovir-emtricitabine for HIV Non-occupational Post-exposure Prophylaxis
Acronym: dPEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrew Carr (Other)
Collaborators: ViiV Healthcare Australia Pty. Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Andrew Carr, Head Clinical research Program, St Vincent's Hospital
Organization: St Vincent's Hospital, Sydney (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2.0 dated 23 June 2014; 201047 (Other Grant/Funding Number: ViiV Healthcare Australia Pty. Ltd)
Record Dates: First submitted 2014-06-23; First posted 2014-08-07 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dolutegravir 50mg with co-formulated emtricitabine-tenofovir (Experimental): One-hundred eligible participants will receive dolutegravir (1 x 50mg tablet) with co-formulated emtricitabine-tenofovir (1 tablet) once daily for 28 days
  Interventions: Drug: dolutegravir 50 mg (one tablet daily); Drug: emtricitabine-tenofovir 300/200 mg (one tablet daily)

INTERVENTIONS:
Drug: dolutegravir 50 mg (one tablet daily)
Drug: emtricitabine-tenofovir 300/200 mg (one tablet daily)

SUMMARY:
This study aims to describe the proportion of participants with non-occupational post-exposure prophylaxis (NPEP) failure, defined as NPEP non-completion (including loss to follow-up) at week 4 or primary HIV infection at week 4 or 12, excluding those participants who should and do cease study drug because:

1. The participant is found to be HIV-infected (study drugs will be ceased until the genotype of the infecting strain is determined)
2. The source is found to be HIV-uninfected

The primary study objectives are:

1. To describe on-drug adherence and regimen completion rates of 28 days of NPEP using dolutegravir (DTG) with co-formulated emtricitabine-tenofovir (FTC-TDF)
2. To describe the safety of 28 days of non-occupational post-exposure prophylaxis (NPEP) using dolutegravir with co-formulated emtricitabine-tenofovir

The study is a multi-site, prospective, open-label, non-randomized trial. One-hundred (100) eligible participants will receive dolutegravir (one tablet) with co-formulated emtricitabine-tenofovir, two tablets, once daily for 28 days based on one of the following exposures:

1. receptive anal intercourse with a source known to be HIV-infected; or
2. receptive anal intercourse with a source of unknown HIV status; or
3. insertive anal intercourse with a source known to be HIV-infected

There will be 7 study visits over a 12-week period. Follow-up post NPEP is for 8 weeks i.e. to week-12 post-exposure. Any participant who is intolerant of dolutegravir will be managed at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Man who has sex with men
2. Age at least 18 years
3. Potential HIV exposure following:

   * receptive anal intercourse with a source known to be HIV-infected; or
   * receptive anal intercourse with a source of unknown HIV status; or
   * insertive anal intercourse with a source known to be HIV-infected
4. Able to provide written, informed consent
5. Able to commit to the study visits

Exclusion Criteria:

1. Non-sexual exposure
2. Exposure occurring during sex between a man and a woman
3. HIV infection diagnosed on baseline testing (antibody, Western blot, proviral DNA) including indeterminate serology consistent with possible primary HIV infection
4. Use of any medication contra-indicated with DTG, FTC or TDF
5. Use of any medication that effects the concentration of dolutegravir and / or concomitant drug including: oxcarbazepine, phenytoin, phenobarbital, carbamazepine, rifampicin, metformin or St. John's wort (St John's wort can be stopped for the 28-day period of NPEP).
6. History or presence of allergy to DTG, FTC, TDF or their components
7. Alanine aminotransferase (ALT) ≥5 times the upper limit of the reference range or ALT ≥3 times and bilirubin ≥1.5 times the upper limit of the reference range
8. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice) or known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
9. Severe hepatic impairment (Class C) as determined by Child-Pugh classification
10. Serum estimated Glomerular Filtration Rate (eGFR) <60 mL/min/BSAc
11. Current therapy for hepatitis B infection
12. Serological evidence of chronic/active hepatitis B
13. Previous OPEP/NPEP containing DTG
14. A participant with a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study, or interfere with the participant's participation for the full duration of the study
15. Unable to complete study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | twelve (12) weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - St Vincent's Hospital Centre for Applied Medical Research, Darlinghurst, New South Wales
  - Sydney Sexual Health Centre, Sydney, New South Wales
  - Clinic 16, Royal North Shore Hospital, Sydney, New South Wales
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Alfred Hospital, Melbourne, Victoria